CLINICAL TRIAL: NCT04694664
Title: Vaccine Confidence Among Pregnant Women and Mothers During the COVID-19 Pandemic
Brief Title: COVID-19 Vaccine Confidence Among Pregnant Women and Mothers
Acronym: VCCOVID
Status: Completed | Type: Observational
Sponsor: Pregistry (Industry)
Collaborators: Harvard School of Public Health (HSPH) (Other)
Responsible Party: Sponsor
Other Study IDs: 0003
Record Dates: First submitted 2020-11-01; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Pregnancy Related; Mothers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnant Women: Pregnant women who are 18 years of age or older.
  Interventions: Other: This is an online survey with no intervention.
- Post-partum women: Women who have at least one child younger than 18 years of age.
  Interventions: Other: This is an online survey with no intervention.

INTERVENTIONS:
Other: This is an online survey with no intervention. — As this is an online survey about health and wellbeing, there is no intervention.

SUMMARY:
The purpose of this study is to assess the level of vaccine confidence and influencers among pregnant women and mothers of school-aged children during the COVID-19 pandemic.

DETAILED DESCRIPTION:
The WHO has listed "vaccine hesitancy" as one of the top threats to global health.

The COVID-19 pandemic has triggered the need to vaccinate worldwide as soon as a safe and efficacious vaccine becomes available. However preliminary data show that, on average, only 50% to 66% of US adults would be willing to receive COVID-19 vaccination when it becomes available, a percentage lower than what is required for herd immunity to control the pandemic. Furthermore, there is a pressing need to vaccinate children to reopen schools and keeping them safe, as well as to immunize pregnant women through vaccination programs since they constitute a vulnerable population. Vaccine confidence among pregnant women and mothers of school-aged children during the period of COVID-19 pandemic is unknown, leading to an important gap of knowledge that may hinder the upcoming global COVID-19 vaccination scale-up effort. It is therefore of critical importance to assess the level of vaccine confidence and influencers among pregnant women and mothers of school-aged children during the COVID-19 pandemic.

The international nature of the proposed survey will allow the evaluation of vaccine confidence and its influencers among pregnant women and mothers of school-aged children on a global level. Therefore, social and geographic characteristics from different countries and cultures will be available for comparison. The resulting knowledge will be relevant to a large percentage of the world's population. Any country in the world can participate.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women or women who have at least one child younger than 18 years of age. Able to give electronic informed consent

Exclusion Criteria:

* <18 years of age

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Persons assigned gender female at birth.
Study Population: Pregnant women or women who have at least one child younger than 18 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 18000 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Percentage of acceptance of a COVID-19 vaccine | up to 2 months
  This outcome will evaluate the hesitancy or acceptance to a COVID-19 vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Julia Wu, SD, MS, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (1):
- Pregistry, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No